CLINICAL TRIAL: NCT02762669
Title: Recovery of Oxytocin Responsiveness in Pregnant Human Myometrial Explants After Oxytocin-Induced Desensitization: an In-vitro Analysis of Oxytocin Receptor Expression and Signaling
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-05
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2024-08-27 (Actual); Status verified 2024-03

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Oxytocin desensitization
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Control (no oxytocin) + No recovery (No Intervention): A control experiment will be undertaken in which the myometrial explants will be exposed to PSS for 2-hours without any oxytocin. No recovery time.
- Continuous oxytocin + No recovery (Active Comparator): 10-5M oxytocin for 2 hours. No recovery time.
  Interventions: Drug: Oxytocin
- Continuous oxytocin + 30 minute recovery (Active Comparator): 10-5M oxytocin for 2 hours. After 2 hours, the solution will be drained from the organ baths, and any residual solution will be removed by washing three times with PSS. Following this, the strip will be exposed to PSS for 30 minutes.
  Interventions: Drug: Oxytocin
- Continuous oxytocin + 60 minute recovery (Active Comparator): 10-5M oxytocin for 2 hours. After 2 hours, the solution will be drained from the organ baths, and any residual solution will be removed by washing three times with PSS. Following this, the strip will be exposed to PSS for 60 minutes.
  Interventions: Drug: Oxytocin
- Control (no oxytocin) + No recovery + 10-7 oxytocin (Active Comparator): A second control experiment will be undertaken in which the myometrial explants will be exposed to PSS for 2-hours without any oxytocin. After 2 hours, the solution will be drained from the organ baths, and replaced with fresh PSS. Following this, the strip will be exposed to 10-7 oxytocin for 10 minutes.
  Interventions: Drug: Oxytocin
- Continuous oxytocin + No recovery + 10-7 oxytocin (Active Comparator): 10-5M oxytocin for 2 hours. After 2 hours, the solution will be drained from the organ baths, and any residual solution will be removed by washing three times with PSS. Following this, the strip will be exposed to 10-7 oxytocin for 10 minutes.
  Interventions: Drug: Oxytocin
- Continuous oxytocin + 30 minute recovery + 10-7 oxytocin (Active Comparator): 10-5M oxytocin for 2 hours. After 2 hours, the solution will be drained from the organ baths, and any residual solution will be removed by washing three times with PSS. Following this, the strip will be exposed to PSS for 30 minutes. The strip will then be exposed to 10-7 oxytocin for 10 minutes.
  Interventions: Drug: Oxytocin
- Continuous oxytocin + 60 minute recovery + 10-7 oxytocin (Active Comparator): 10-5M oxytocin for 2 hours. After 2 hours, the solution will be drained from the organ baths, and any residual solution will be removed by washing three times with PSS. Following this, the strip will be exposed to PSS for 60 minutes. The strip will then be exposed to 10-7 oxytocin for 10 minutes.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 10-7mol/L to 10-5mol/L
  Other Names: pitocin
  Arms: Continuous oxytocin + 30 minute recovery; Continuous oxytocin + 30 minute recovery + 10-7 oxytocin; Continuous oxytocin + 60 minute recovery; Continuous oxytocin + 60 minute recovery + 10-7 oxytocin; Continuous oxytocin + No recovery; Continuous oxytocin + No recovery + 10-7 oxytocin; Control (no oxytocin) + No recovery + 10-7 oxytocin

SUMMARY:
Postpartum hemorrhage (PPH) is a leading cause of maternal mortality and morbidity worldwide, and is caused most commonly by poor uterine muscle contraction after delivery of the baby and placenta. The first line agent used in the prevention and treatment of PPH is oxytocin, which acts by binding with the oxytocin receptor (OTR) found on myometrial cells to cause uterine contraction.

Oxytocin is also used for the augmentation of labor when spontaneous labor has been deemed ineffective. It is administered intravenously at progressively higher doses, until effective contractions are achieved and vaginal delivery results. However, if augmentation is determined to have failed, a Cesarean delivery (CD) is performed.

One of the potential problems with oxytocin use during delivery is that it loses its effectiveness if the uterus has previously been pre-exposed to its high doses and/or for a prolonged duration during labor. This phenomenon is termed OTR desensitization, and can result in the attenuation of myometrial contractility induced by subsequent oxytocin administration, as well as PPH due to poor uterine tone. Furthermore, oxytocin can produce potentially fatal maternal hemodynamic adverse effects when administered at high doses, so it is advantageous to be able to use as low a dose as possible to obtain good uterine muscle tone.

The objective of this study is to get a better understanding of the signaling pathways governing desensitization, resensitization and contractility in pregnant human myometrium. The investigators wish to investigate the effects of increasing recovery period on the expression patterns of the OTR and its signaling pathways in desensitized pregnant human myometrium.

This study will help shed light on the molecular mechanisms responsible for desensitization and oxytocin-induced myometrial contractility, and will provide some insight into potential therapeutic targets to reduce the incidence of PPH and complications associated with using increasing concentrations of oxytocin.

The hypothesis is that the expression and phosphorylation patterns of the OTR and downstream proteins will be altered in desensitized myometrium, and that these patterns will change with increasing rest periods and re-exposure to oxytocin.

DETAILED DESCRIPTION:
Clinically, women who require augmentation of labor are at increased risk of PPH due to their greater exposure to oxytocin in both duration and dose through exogenous administration, presumably mediated by OTR desensitization. In current practice, upon diagnosis of failure to progress during labor augmentation, oxytocin administration is discontinued, and as long as there is no indication for immediate delivery, there is a variable duration to proceed to CD. Due to the high likelihood of OTR desensitization in this patient population, it would be clinically relevant to determine the molecular mechanisms underlying this action.

A recent study from the investigators' group, looking at the rest time required for recovery and resensitization of the OTR following desensitization, showed that there were no improvements in oxytocin-induced myometrial contractility after either a 30, 60 or 90 minute rest period. The reason for why resensitization does not occur remains unknown, but a possible explanation is that the OTRs undergo structural and functional changes during desensitization that prohibit their recovery.

The investigators propose to use our previously established in-vitro model of labour augmentation and OTR desensitization (using pregnant human myometrium and an isometric tension recording device) to investigate the molecular mechanisms governing OTR desensitization and resensitization after stopping administration of oxytocin. Investigation of the signaling pathways responsible for these processes, as well as for oxytocin-induced contractions in a controlled in-vitro system will aid in the understanding of the kinetics of the OTR-oxytocin system and provide insight into potential pharmacotherapeutic targets to reduce the incidence of PPH.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary Cesarean delivery or first repeat Cesarean delivery

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients who had previous uterine surgery or more than one previous Cesarean delivery
* Patients with any condition predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, bleeding diathesis, chorioamnionitis, or a previous history of postpartum bleeding
* Emergency Cesarean section in labor
* Patients on medications that could affect myometrial contractility, such as nifedipine, labetolol or magnesium sulphate.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Oxytocin receptor (OTR) protein expression and localization | 24 hours
  Western blotting will be performed to detect expression levels of the OTR protein and its localization within the plasma membrane, cytoplasmic or nuclear cell fractions.

SECONDARY OUTCOMES:
Oxytocin receptor (OTR) phosphorylation patterns | 24 hours
  Proximity assays will be used to detect OTR phosphorylation patterns, by looking at the extent of OTR-β-arrestin binding.
Protein expression levels of PLC, MEK5 and ERK5 | 24 hours
  Western blotting will be performed to detect protein expression levels of PLC, MEK5 and ERK5

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No